CLINICAL TRIAL: NCT06778018
Title: Effects of Lotus Seed (Nelumbo Nucifera) on the Nutritional, Electrophysiological and Immunomodulatory Outcomes in Patients With Diabetic Sensorimotor Polyneuropathy
Brief Title: Nutritional Outcomes of Lotus Seed (Nelumbo Nucifera) on Diabetic Sensorimotor Polyneuropathy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: REC/RCR&AHS/24/1301
Record Dates: First submitted 2024-12-20; First posted 2025-01-16 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Diabetes Mellitus, Type 2; Diabetic Nephropathies
Keywords: Diabetic Sensorimotor Polyneuropathy; Lotus Seed; Electrophysiological; Neuroprotective; Type 2 Diabetes; Nutritional
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetic Nephropathies

STUDY DESIGN:
Intervention Model Description: it will be a randomized controlled trial in which non probability convenient sampling will be used. Two groups of 40 and above age will be formed in which participants will be randomly divided. Group A (Control group) will receive the standard antidiabetic regimen along with a placebo capsules (Starch) at the dose rate of 200mg/kg. , while Group B (Treatment group) will receive the same antidiabetic regimen supplemented with Lotus Seed capsules at a dose of 200 mg/kg.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Control group) (Placebo Comparator): This group will receive the placebo treatment (starch) 200 mg/kg capsules. Baseline assessments will be conducted before the intervention, followed by health evaluations at 6 months (end of intervention), 9 months, and 12 months (follow-up assessments). Comprehensive health assessments will include nutritional status (BMI, dietary intake), biochemical markers (HbA1c, lipid profile, liver, and kidney function), and electrophysiological tests (Neuropathy Disability Score and immune-modulatory response). The data collected will be analyzed using SPSS version 25, allowing for comparisons between pre- and post-intervention outcomes in both groups.
  Interventions: Dietary Supplement: Placebo
- Group B (Treatment group) (Experimental): This group will receive the intervention treatment 200 mg/kg Lotus Seed capsules. Baseline assessments will be conducted before the intervention, followed by health evaluations at 6 months (end of intervention), 9 months, and 12 months (follow-up assessments). Comprehensive health assessments will include nutritional status (BMI, dietary intake), biochemical markers (HbA1c, lipid profile, liver, and kidney function), and electrophysiological tests (Neuropathy Disability Score and immune-modulatory response). The data collected will be analyzed using SPSS version 25, allowing for comparisons between pre- and post-intervention outcomes in both groups.
  Interventions: Dietary Supplement: Lotus Seed

INTERVENTIONS:
Dietary Supplement: Lotus Seed — Regimen supplemented with 200 mg/kg of Lotus Seed capsules for 12-month randomized controlled trial.
  Arms: Group B (Treatment group)
Dietary Supplement: Placebo — Regimen supplemented with 200 mg/kg of Starch capsules for 12-month randomized controlled trial.
  Arms: Group A (Control group)

SUMMARY:
The study focuses on Diabetic Sensorimotor Polyneuropathy (DSPN), a common complication of type 1 and type 2 diabetes caused by hyperglycemia-induced nerve damage, leading to pain, numbness, and motor dysfunction in the limbs. It also affects the digestive system, urinary tract, and cardiovascular health, often resulting in diabetic foot ulcers, amputations, and reduced quality of life. Current management involves glycemic control, pain relief, and complication prevention. Recent research highlights the neuroprotective potential of Lotus (Nelumbo nucifera) in promoting axonal regeneration, suppressing apoptosis, and enhancing motor function recovery. This randomized controlled trial will investigate the anti-diabetic effects of Lotus Seed in type 2 diabetes patients at a private hospital in Lahore, Pakistan, over 12 months. Participants will be divided into a control group receiving a standard antidiabetic regimen with placebo capsules and a treatment group receiving 200 mg/kg of Lotus Seed capsules alongside the antidiabetic regimen. Baseline characteristics and post-intervention changes will be assessed through nutritional impact (BMI, dietary intake), serum biochemical tests (HbA1c, lipid profile, liver, and renal function), and electrophysiological tests (Neuropathy Disability Score and immune-modulatory tests). Data collection will occur at baseline, 6 months (end of intervention), and follow-ups at 9 and 12 months. SPSS version 25 will be used for statistical analysis to evaluate the potential of Lotus Seed as a functional food for managing DSPN and improving health outcomes in diabetic patients.

DETAILED DESCRIPTION:
The research project aims to investigate the therapeutic impact of Lotus Seed (Nelumbo nucifera) on Diabetic Sensorimotor Polyneuropathy (DSPN), a common complication observed in patients with type 1 and type 2 diabetes. DSPN is caused by chronic hyperglycemia, which leads to the degeneration of sensory and motor nerves, particularly the long peripheral nerves that extend to the arms, hands, legs, and feet. This damage results in pain, tingling, numbness, and loss of motor control. Additionally, DSPN can affect the functioning of the digestive system, urinary tract, blood vessels, and cardiovascular system. Over time, it serves as a precursor to more severe complications such as non-healing diabetic wounds, infections, diabetic foot ulcers, amputations, and, in extreme cases, death. The resulting neurological dysfunctions significantly reduce the quality of life for diabetic patients.

Conventional management of DSPN emphasizes glycemic control, symptom relief, and the prevention of long-term complications. Treatment options typically include medications for pain relief, such as neuropathic pain medications, alongside lifestyle changes and regular health monitoring. However, emerging research suggests that functional foods with neuroprotective properties, such as Lotus Seed, may offer an alternative or complementary approach. Histological studies indicate that Lotus exhibits neuroprotective and regenerative effects on nerve cells by inhibiting cellular apoptosis, especially during the acute injury phase. It has also been found to support axonal regeneration, reduce axonal dieback, and enhance motor function recovery. Additionally, Lotus overexpression has been shown to improve neuronal plasticity in the brainstem and cervical spinal cord after stroke, demonstrating its potential for future therapeutic applications in nerve-related disorders.

This study will be a 12-month randomized controlled trial (RCT) conducted at a private hospital in Lahore, Pakistan, targeting patients with a confirmed diagnosis of type 2 diabetes mellitus (T2DM). The participants will be randomly assigned to one of two groups. Group A (Control group) will receive the standard antidiabetic regimen along with a placebo capsule, while Group B (Treatment group) will receive the same antidiabetic regimen supplemented with Lotus Seed capsules at a dose of 200 mg/kg. The intervention period will last for 6 months, followed by two post-intervention follow-ups at 9 and 12 months to monitor the sustainability of the treatment effects. Before enrollment, all participants will provide informed consent, and their baseline health status will be assessed through comprehensive testing.

The key parameters to be evaluated include both nutritional, biochemical, and electrophysiological markers. Nutritional impact will be measured through anthropometric indices (such as Body Mass Index), dietary intake assessments, and changes in overall nutritional status. Serum biochemical tests will analyze metabolic markers, including glycemic parameters (HbA1c), lipid profile, liver function, and renal function. Neurological assessments will include the Neuropathy Disability Score and an evaluation of immune-modulatory responses to track changes in nerve function. These tests will be conducted at four time points: baseline (pre-intervention), 6 months (end of intervention), 9 months (follow-up), and 12 months (final follow-up).

All collected data will be analyzed using SPSS version 25. Statistical analysis will focus on comparing changes in health outcomes between the control and treatment groups to determine the impact of Lotus Seed supplementation on DSPN management. This research aims to establish evidence for the use of Lotus Seed as a functional food that can complement standard medical treatment, promoting nerve regeneration, improving metabolic parameters, and enhancing the overall health and well-being of patients with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Participants who have been clinically diagnosed with T2DM (Type 2 Diabetes Mellitus).
* Participants who have been clinically diagnosed with neuropathy symptoms for at least 1 year.
* Both male and female participants.
* Participants aged 40 years and older.
* Participants capable of understanding basic instructions, either independently or with assistance from their family.

Exclusion Criteria:

* Individuals with a clinical diagnosis of cardiovascular conditions.
* Cancer patients will be excluded from the study.
* Individuals diagnosed with rheumatoid arthritis.
* Individuals with a urinary tract infection.
* Individuals diagnosed with psychological disorders.
* Pregnant or breastfeeding women.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-12-10 (Actual); Primary Completion 2025-12-10 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Body Mass Index (BMI) | 12 months
  The Body Mass Index (BMI) will be calculated based on an individual's height and weight. Height will be measured using a stadiometer, and weight will be assessed with a weighing scale. BMI will be derived by dividing the weight in kilograms by the square of the height in meters. The classification thresholds established by the World Health Organization (WHO) will be utilized for interpretation.
HbA1c | 12 months
  The HbA1c level of 6.5% will be measured by drawing blood from the individuals, followed by analysis to detect the presence of diabetes.
Lipid Profile | 12 months
  A blood lipid profile will be collected from the individuals, and the analysis will be performed at the Private Hospital. The lipid profile will assess total cholesterol, very low-density lipoprotein (VLDL), low-density lipoprotein (LDL), high-density lipoprotein (HDL), and triglyceride levels.
Alanine Transaminase (ALT) | 12 months
  Liver function tests will be performed by collecting blood from the individuals, and the analysis will take place at the Private Hospital. These tests will measure alanine transaminase (ALT). The tests will be conducted using semi-automatic or fully automated machines that operate on photometric principles.
Liver Function Test-aspartate transaminase (AST) | 12 months
  Liver function tests will be performed by collecting blood from the individuals, and the analysis will take place at the Private Hospital. These tests will measure aspartate transaminase (AST). The tests will be conducted using semi-automatic or fully automated machines that operate on photometric principles.
Liver Function Test-alkaline phosphatase (ALP) | 12 months
  Liver function tests will be performed by collecting blood from the individuals, and the analysis will take place at the Private Hospital. These tests will measure alkaline phosphatase (ALP). The tests will be conducted using semi-automatic or fully automated machines that operate on photometric principles.
Liver Function Test-gamma-glutamyl transferase (GGT) | 12 months
  Liver function tests will be performed by collecting blood from the individuals, and the analysis will take place at the Private Hospital. These tests will measure gamma-glutamyl transferase (GGT). The tests will be conducted using semi-automatic or fully automated machines that operate on photometric principles.
Liver Function Test-serum bilirubin | 12 months
  Liver function tests will be performed by collecting blood from the individuals, and the analysis will take place at the Private Hospital. These tests will measure serum bilirubin. The tests will be conducted using semi-automatic or fully automated machines that operate on photometric principles.
Liver Function Test-prothrombin time (PT) | 12 months
  Liver function tests will be performed by collecting blood from the individuals, and the analysis will take place at the Private Hospital. These tests will measure prothrombin time (PT). The tests will be conducted using semi-automatic or fully automated machines that operate on photometric principles.
Liver Function Test-international normalized ratio (INR) | 12 months
  Liver function tests will be performed by collecting blood from the individuals, and the analysis will take place at the Private Hospital. These tests will measure international normalized ratio (INR). The tests will be conducted using semi-automatic or fully automated machines that operate on photometric principles.
Liver Function Test-total protein | 12 months
  Liver function tests will be performed by collecting blood from the individuals, and the analysis will take place at the Private Hospital. These tests will measure total protein. The tests will be conducted using semi-automatic or fully automated machines that operate on photometric principles.
Liver Function Test-albumin | 12 months
  Liver function tests will be performed by collecting blood from the individuals, and the analysis will take place at the Private Hospital. These tests will measure albumin. The tests will be conducted using semi-automatic or fully automated machines that operate on photometric principles.
Renal Function Test-serum creatinine | 12 months
  Renal function tests will be carried out by drawing blood from the individuals, and the analysis will be conducted at a private hospital. These tests will assess various markers of kidney function like serum creatinine. Based on photometric principles, the tests will be performed using semi-automatic or fully automated analyzers.
Renal Function Test-blood urea nitrogen (BUN) | 12 months
  Renal function tests will be carried out by drawing blood from the individuals, and the analysis will be conducted at a private hospital. These tests will assess various markers of kidney function like blood urea nitrogen (BUN). Based on photometric principles, the tests will be performed using semi-automatic or fully automated analyzers.
Renal Function Test- glomerular filtration rate (GFR) | 12 months
  Renal function tests will be carried out by drawing blood from the individuals, and the analysis will be conducted at a private hospital. These tests will assess various markers of kidney function like glomerular filtration rate (GFR). Based on photometric principles, the tests will be performed using semi-automatic or fully automated analyzers.
Renal Function Test-electrolytes such as sodium, potassium, and chloride | 12 months
  Renal function tests will be carried out by drawing blood from the individuals, and the analysis will be conducted at a private hospital. These tests will assess various markers of kidney function like electrolytes such as sodium, potassium, and chloride. Based on photometric principles, the tests will be performed using semi-automatic or fully automated analyzers.
Neuropathy disability score (NDS) | 12 months
  The Neuropathy Disability Score (NDS) is a widely used clinical tool to evaluate signs of neuropathy. This assessment focuses on four key signs of neuropathy: ankle reflex, vibration sensation, pinprick sensation, and temperature perception, all tested on both sides of the largest toes. The total possible score is 10, with scores above 6 typically indicating an abnormal result.
Cell mediated Response CD4, CD3 and CD8. | 12 months
  The patient's immune response will be assessed by measuring CD4, CD3, and CD8 levels at the Private Hospital. CD4 cells are the predominant T cells in healthy individuals and play a crucial role in assisting B cells with antibody production and enhancing immune reactions to antigens. CD4 cell count is often used as an indicator of immune suppression, with lower levels suggesting a gradual decline in immune function.
Immunoglobulins | 12 months
  The patient's immune function will be assessed by measuring the levels of IgA, IgG, and IgM antibodies. These antibodies are proteins that the immune system generates to combat harmful microorganisms such as bacteria and viruses. The immunoglobulin test can help determine if there are any issues with the immune system, as certain conditions may lead to an imbalance in antibody production. IgM antibodies are the first to be produced after the body is exposed to pathogens, providing temporary defense until other antibodies are formed. These antibodies are present in the blood and lymph. IgG antibodies play a key role in fighting bacterial and viral infections, while IgA antibodies protect the respiratory and digestive systems.

CONTACTS AND LOCATIONS:
Overall Officials: Moha Akram Khan, PhD*, Principal Investigator — Riphah International University
Locations (1):
- Riphah international university, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhu J, Hu Z, Luo Y, Liu Y, Luo W, Du X, Luo Z, Hu J, Peng S. Diabetic peripheral neuropathy: pathogenetic mechanisms and treatment. Front Endocrinol (Lausanne). 2024 Jan 9;14:1265372. doi: 10.3389/fendo.2023.1265372. eCollection 2023. PMID 38264279